CLINICAL TRIAL: NCT03069261
Title: Intraoperative Indocyanine Green Laser (ICG) Angiography; Evaluation of Postoperative Outcomes for Breast Reconstruction With Autologous Tissue Flaps
Brief Title: Intraoperative Indocyanine Green Laser Angiography; Postoperative Outcomes for Autologous Tissue Flaps
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: ICG-angiography
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: Breast reconstruction; Autologous tissue flaps; Indocyanine green angiography; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention - ICG angiography: ICG-angiography was used intraoperatively after placement of the flap at the recipient cite, evaluating the viability and perfusion of the flap. Poor perfused areas were excised
  Interventions: Device: Indocyanine green angiography
- Control - clinical assessment: A control group receiving identical operations but without ICG-angiography evaluation.

INTERVENTIONS:
Device: Indocyanine green angiography
  Groups: Intervention - ICG angiography

SUMMARY:
The purpose of this study is to identify and compare complication rates between autologous breast reconstruction techniques with and without the inclusion on intraoperative indocyanine green (ICG) angiography.

DETAILED DESCRIPTION:
ICG-angiography is a real-time visualization of tissue perfusion using intravenous fluorescence. It allows the surgeon a tool for intraoperatively assessment of tissue perfusion of the autologous flap, providing a basis for trimming of hypo perfused areas. The study evaluates the effect of inclusion of this technique by examine postoperative outcomes retrospectively. This is done by differentiation between major and minor complications to evaluate the greatest gains of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients over the age of 18 years
* Deemed suitable for breast reconstruction with the latissimus dorsi (LD) myocutaneous flap, muscle sparring LD flap or transverse rectus abdominal muscle (TRAM) flap

Exclusion Criteria:

* Patients with recurrence of breast cancer
* Smoking 4 weeks prior of operation
* Not able to read and understand Danish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who underwent immediate or delayed, pedicle autologous flap breast reconstruction between 2012 and 2016 were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Major complications | Measured at 6 months followup.
  Major complications included necrosis of most of the flap (2/3), total flap loss and surgical evacuated hematoma.

SECONDARY OUTCOMES:
Minor complications | Measured from day 0 with 6 months followup
  A minor complication included clinical sign of infection, prolonged wound healing (defined as prolonged healing time requiring dressing changes assisted by health personnel), fat necrosis and skin necrosis.
Timing of reconstruction | Measured from day 0 with 6 months followup
  Comparison of the timing of the reconstruction with the complication rate, comparing immediate reconstructions with delayed reconstructions.